CLINICAL TRIAL: NCT04538430
Title: Medial Branch Peripheral Nerve Stimulation for Refractory Axial Back Pain
Brief Title: Peripheral Nerve Stimulation for Back
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 and other factors this study was terminated early and the patients currently enrolled are being used as a small pilot study.
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Zack McCormick, Zachary McCormick, MD FAAPMR, Associate Professor, Director of Clinical Spine Research, Director of Interventional Spine and Musculoskeletal Medicine Fellowship, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 127414
Record Dates: First submitted 2020-08-28; First posted 2020-09-04 (Actual); Results first posted 2022-11-23 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Back Pain
Keywords: Axial Low Back Pain; Peripheral Nerve Stimulation; Medial Branches
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Axial Low Back Pain (Other): Patient diagnosed with axial low back pain not responding to conservative measures and no symptoms of radiculopathy, that is scheduled to have a SPRINT percutaneous peripheral nerve stimulator placed as standard of care.
  Interventions: Device: SPRINT percutaneous peripheral nerve stimulator placed

INTERVENTIONS:
Device: SPRINT percutaneous peripheral nerve stimulator placed — Placement of a SPRINT percutaneous peripheral nerve stimulator targeting the bilateral medial branches at the suspected level of pain generation. This procedure is done as standard of care.

SUMMARY:
To assess changes in pain, physical function, health-related quality of life, and cost-effectiveness in patients with low back pain, without symptoms of radiculopathy, that have not responded to conservative or traditional interventional measures and are having a SPRINT percutaneous peripheral nerve stimulator placed as standard of care. Patients will be assessed periodically (by questionnaire) after the placement of the SPRINT, FDA approved 60 day, percutaneous peripheral nerve stimulator, targeting the bilateral medial branches at the suspected level of pain generation. Neither the manufacturer nor the FDA are involved or will have access to data from this study.

DETAILED DESCRIPTION:
Low back pain is one of a few conditions which affects all individuals through the lifespan. The etiology of low back pain is multifactorial and in many cases self-limiting, however it also is the leading cause for working age adults to be disabled with more than $87 billion spent on low back pain disorders in 2013. Listhesis of a vertebral body, chronic compression fractures, lumbar disc herniation, and internal disc disruptions are some primary anatomical abnormalities that can cause back pain and do not have great targeted treatments. that may more common in these younger age groups reaching 39-42% with a predicted probability above 60% until age 50y. While the natural history of back pain suggests most individuals will return to a prior level of function in 3-6 months, there is a high rate of recurrent episodes which can cause short-term disability. Continued back pain can lead to decreased activity levels and accelerate degenerative changes in the disc and facet joints as described by Kirkaldy-Willis.

Current guidelines for treatment of axial low back pain include a 6-12-week course of conservative care including medications, therapy, acupuncture, chiropractic and exercise before an interventional paradigm of injections and/or surgical treatment. For those individuals who do not improve with conservative care and have predominately axial pain, options are limited as success rates from epidural steroid injections and surgery are 50% or less. Other treatments include chymopapain injection, intradiscal electrothermal annuloplasty (IDET), nucleoplasty, methylene blue injection. All of which have 50% or less likelihood of reducing pain more than 50%, although much of this data is from uncontrolled or prospective case-control studies only.

Peripheral Nerve Stimulation (PNS) recently gained FDA approval as an interventional treatment of chronic back pain. PNS involves a minimally invasive percutaneous microelectrode connected to an external impulse generator that adheres to the skin for up to 60 days and then the entire system is removed. It is theorized that the neuromodulatory effects of PNS interrupts the chronic pain cycle and allowing healthy recovery of afferent signaling and limiting and perhaps reversing the maladaptive cortical plasticity involved in chronic pain. There have been two prospective cohort studies published this year, both of which showed meaningful clinical improvement in pain and function scores. One of these studies (Cohen et al.) showed that more than 50% of the patients had greater than 50% improvement in pain at one year after undergoing 2 months of implanted PNS treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years of age at day of enrollment.
2. Clinical diagnosis of refractory low back pain for >3 months.
3. Magnetic resonance imaging pathology consistent with clinical symptoms/signs at one or two levels.
4. Back pain of at least 4/10 or higher using the Numerical Rating Scale (NRS).
5. Pain duration of more than 12 weeks despite trial of conservative therapy (medications, physical therapy, or chiropractic care) for 2 months.

Exclusion Criteria:

1. Refusal to participate, provide consent, or provide follow-up information for the 24-month duration of the study.
2. Contraindications to medial branch targeted PNS (active infection, bleeding disorders, current anticoagulant or antiplatelet medication use, allergy to iodinated contrast, penicillin or clindamycin and pregnancy or breastfeeding).
3. More than 2 levels of clinical proven pain.
4. Active moderate to severe lumbar radiculopathy.
5. Intradural disc herniation.
6. Spinal fracture of posterior elements within the past 6 months.
7. Steroid injection in the spine within the last 30 days.
8. Any intradiscal injection other than contrast dye or anesthetic in the last 30 days.
9. Prior fusion at level considered to be the source of the pain.
10. Prior lumbar spine surgery within the last 6 months.
11. AP diameter of spinal canal less than or equal to 9mm at level to be treated.
12. Severe uncontrolled medical condition.
13. Severe psychological illness.
14. History of Inflammatory arthritis.
15. Malignancy within past 5 years except basal cell or squamous cell skin cancer.
16. Current use of equal to greater than 45mg morphine-equivalent per day of opioid use.
17. A history of alcohol or drug abuse within past 5 years.
18. Use of any investigational drug within past 30 days.
19. Severe anaphylactic/anaphylactoid reaction to any medications used.
20. Pending litigation involving subject's back pain.
21. No insurance coverage for any subsequent tests or procedures.
22. Inability or unwillingness to continue rehabilitation protocols.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-09-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah Orthopaedic Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Axial Low Back Pain
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Axial Low Back Pain
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Pain Numeric Rating Scale (NRS) Response From SPRINT Percutaneous Peripheral Nerve Stimulator
Description: Assessment of Pain Numeric Rating Scale (0-10) response after placement of SPRINT percutaneous peripheral nerve stimulator for chronic low back pain. 0 being no pain and 10 being the worst pain.
Time Frame: 2 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Axial Low Back Pain
Number analyzed (Participants) | 7
score on a scale | 3.17 [0 to 10]

ADVERSE EVENTS:
Time Frame: up to 21 months.
Description: No adverse events were reported during the duration of this study.
Arm/Group | Axial Low Back Pain
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/30/NCT04538430/Prot_SAP_000.pdf